CLINICAL TRIAL: NCT01946360
Title: Role of 13C Methacetin Breath Test in Predicting Prognosis Among Patients With Acute or Acute on Chronic Liver Failure (ACLF).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ILBS-ACLF-MBT-01
Record Dates: First submitted 2013-08-22; First posted 2013-09-19 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Acute Liver Failure; Acute on Chronic Liver Failure
MeSH Terms: conditions — Liver Failure, Acute; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACLF and Acute Liver Failure (ALF).. (No Intervention): Methacetin Breath Test will be done on Day 0,7,14,28 in Acute on Chronic Liver Failure (ACLF)and on day 0,1,3,7 in Acute Liver failure (ALF).
  Interventions: Device: Methacetin Breath Test in ACLF and ALF patients

INTERVENTIONS:
Device: Methacetin Breath Test in ACLF and ALF patients — Methacetin Breath Test will be done on Day 0,7,14,28 in Acute on Chronic Liver Failure (ACLF)and on day 0,1,3,7 in Acute Liver failure (ALF).

SUMMARY:
Blood will be collected after venepuncture from all patients for complete blood counts, Serum bilirubin (direct and indirect), aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma glutamyl transferase, prothrombin time and INR, urea, creatinine, sodium, potassium, serum total protein and albumin, within 24 hours after admission and twice a week there after or as and when needed.

Time line for blood tests and evaluation of clinical parameters & 13C-MBT

For ALF patients:

On days 0, 1, 3, and 7

For ACLF patients:

On days 0, 7 (week 1), 14(week 2), 28 (weeks 4)

Blood tests would include:

Serum bilirubin (total and direct), aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyltransferase, Serum proteins (total and albumin), prothrombin time & international normalized ratio (INR), Serum urea and creatinine, serum electrolytes, arterial ammonia and arterial blood gas analysis.

ELIGIBILITY:
Inclusion Criteria:

- All patients presenting with acute liver failure and acute on chronic liver failure (between 18 - 70 years of age) to Institute of Liver & Biliary Sciences (ILBS), New Delhi, India.

Exclusion Criteria:

1. Patients with significant co-morbid illnesses such as cardiovascular or respiratory or intrinsic renal diseases which by themselves may have a bearing on the outcome.
2. Patients with previous intestinal bypass surgery for morbid obesity
3. Patients with extensive small bowel resection
4. Patients currently receiving total parenteral nutrition
5. Pregnant women
6. Patients with history of allergy to paracetamol
7. Patients on steroids or anti-fungal agents
8. Patients in encephalopathy
9. Patients unwilling to participate in the protocol
10. Patients on medications which can alter the activity of CYP 1A2 enzymes such as corticosteroids, amiodarone, tetracycline, niacin, valproic acid, methotrexate, stavudine and zidovudine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Survival or Transplantation for Acute Liver Failure (ALF). | 2 years

SECONDARY OUTCOMES:
Mortality or Transplantation for Acute on Chronic Liver Failure (ACLF) patients. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ashok Choudhary, DM, Principal Investigator — Institute of Liver & Biliary Sciences.
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India